CLINICAL TRIAL: NCT02210494
Title: Phase 1 Study of Safety of Secretrol® in the Short-term Management of Patients Undergoing Endoscopic Mucosal Resection (EMR)
Brief Title: Safety of Secretrol® in the Short-term Management of Patients Undergoing Endoscopic Mucosal Resection (EMR)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Effexus Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP202
Record Dates: First submitted 2014-08-01; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: EMR Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Secretrol (Experimental)
  Interventions: Drug: Secretrol

INTERVENTIONS:
Drug: Secretrol

SUMMARY:
Evaluate the safety of Secretrol® in patients undergoing endoscopic mucosal resection for early adenocarcinoma of the esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Category 4-high-grade intraepithelial neoplasia
* Ages 18 or older
* signed Informed Consent Form
* signed Health Insurance Portability and Accountability Act (HIPAA) Authorization Form

Exclusion Criteria:

* Clinically relevant data suggesting an unknown disease and requiring further evaluation by the Primary Investigator.
* Patients with renal failure or organ transplants.
* Patients who have known allergic reactions to Proton Pump Inhibitors (PPI).
* Participation in another study that would interfere with study endpoints within 30 days prior to screening.
* Previous enrollment into the current study.
* Patient is the Investigator, his family member or employee at the investigational site.
* Patient known or suspected to be involved in alcohol or drug abuse.
* Known or suspected history of non-compliance with medications.
* Inability to follow the procedures of the study (e.g., due to language problems, psychological disorders)
* Patients receiving prohibited concomitant medications including PPIs, H2-blockers, sucralfate, misoprostol.
* Patients receiving prohibited concomitant medications including clopidogrel, ketoconazole, digoxin, diazepam, warfarin, phenytoin, emtricitabine/nelfinavir/tenofovir, atazanavir, citalopram, emtricitabine/rilpivirine/tenofovir, rilpivirine, nelfinavir, tricyclic antidepressants, baclofen, tacrolimus, cyclosporine, cilostazol, disulfiram, methotrexate, voriconazole.
* Pregnancy or intention to become pregnant during the course of study, breast feeding, or unwillingness to use a highly effective means of contraception (oral contraception or intrauterine device).
* Prescription Non-steroidal anti-inflammatory Drug (NSAID) or aspirin use: The patient must be able to stop these meds 1 week prior to screening and during treatment.
* History of upper gastrointestinal surgery, Zollinger-Ellison syndrome, esophageal stricture, peptic stricture, duodenal and ⁄ or gastric ulcer, esophageal motility disorders, Inflammatory Bowel Disease (IBD), AIDS, pancreatitis, malabsorption, severe cardiovascular or pulmonary disease, liver disease, active malignant disease, Scleroderma, diabetes mellitus, autonomic or peripheral neuropathy, myopathy, functional bowel disorder or any underlying disease or medication that might affect the lower esophageal sphincter pressure or increase the acid clearance time.
* Subject unable or unwilling to fully complete all stages of the study.
* Unable to sign informed consent or inability to give fully informed consent due to language problems, psychological disorder or mental deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Adverse effect evaluation | 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Veteran's Administration Medical Center, Kansas City, Missouri, United States